CLINICAL TRIAL: NCT01531725
Title: 6 Months Evaluation of the BIOTRONIK PRO-Kinetic Coronary Stent System
Brief Title: MULTIcentric BElgium/NEtherlands PRO-Kinetic Safety and Efficacy Study
Acronym: MULTIBENE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0601
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: Stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMS implantation (Experimental): Patients meeting the inclusion criteria and none of the exclusion criteria are treated by implanting the study device (the ProKinetic bare metal stent). Since it is a single arm study design, no patients are enrolled to a control arm.
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — Percutaneous coronary intervention
  Other Names: PRO-Kinetic stent system

SUMMARY:
The primary objective of this study is to evaluate safety and efficacy of the BIOTRONIK PRO-Kinetic coronary CoCr-stent in patients with single de novo lesions of native coronary arteries.

DETAILED DESCRIPTION:
The PRO-Kinetic study is a multi-center, prospective, consecutive non-randomized study enrolling 200 patients with single de novo lesions in native coronary arteries meeting the entry criteria. Those who provide informed consent will be enrolled to receive the PRO-Kinetic stent. Telephone follow-up will be performed at 1 month for all enrolled patients. After 6 months 100 patients will have an angiographic follow-up and 100 patients will be checked by telephone again. Additionally, a clinical telephone follow-up will be performed in all patients after 12 months.

This study is designed to yield data on the clinical safety and efficacy of the PRO-Kinetic stent in the coronary artery application. The Target Vessel Failure Rate after 6 months shall be below 18 % (max. 35 Serious Adverse Events and Expedited Events) to show a safety/performance profile that could be considered in the range of the currently available bare metal stent systems

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years old.
* Eligible for percutaneous coronary intervention (PCI).
* Documented stable (Canadian Cardiovascular Society Classification [CCS] 1, 2, 3, or 4) or unstable (Braunwald type I, II, III and A, B or C) angina pectoris, or documented silent ischemia.
* Left ventricular ejection fraction (LVEF) > 30% documented within the last 6 weeks.
* Acceptable candidate for coronary artery bypass graft surgery (CABG).
* Patient understands the study requirements and the treatment procedures and provides written Informed Consent on a form that has been approved the by local Institutional Review Board before any specific test of the study or procedure is performed.
* Willing to comply with all the specified follow-up evaluations.
* Single target vessels to be treated.
* Single target lesion to be treated.
* Target lesion must be completely coverable by one study stent.
* Total target lesion length <20 mm based on a visual estimate.
* RVD of ≥ 2.0 mm to ≤ 5.0 mm based on a visual estimate.
* Target lesion diameter stenosis ≥ 50% and < 100% based on a visual estimate.
* Target lesion has not undergone prior revascularization up to now.
* Target vessel has not undergone prior revascularization within the preceding 6 months.
* Patient has no child bearing potential, is not pregnant, or intends to become pregnant during the study.

Exclusion Criteria:

* Planned treatment with any other PCI device in target vessel except the pre-dilatation balloon.
* MI within 72 hours prior to the index procedure and/or creatine kinase (CK) > 2 times the local laboratory upper limits of normal, measured on the day of the index procedure, associated with elevated MB.
* The patient is in cardiogenic shock.
* Cerebrovascular Accident (CVA) within the past 6 months.
* Acute or chronic renal dysfunction (creatinine > 2.0 mg/dl or > 150 µmol/L).
* Contraindication to ASA or to clopidogrel.
* Known Thrombocytopenia (platelet count 100, 000/mm3).
* Active gastrointestinal (GI) bleeding within the past three months.
* Known allergy to stainless steel or cobalt chromium.
* Any prior true anaphylactic reaction to contrast agents.
* Patient is currently taking colchicine.
* Life expectancy of less than 24 months due to other medical conditions.
* Co-morbid condition(s) that could limit the patient's ability to participate in the study, compliance with follow-up requirements or impact the scientific integrity of the study.
* Currently participating in another investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.
* Left main coronary artery disease (stenosis > 50%), whether protected or unprotected.
* Target lesion site is ostial (within 3.0 mm of vessel origin).
* Target lesion and/or target vessel proximal to the target lesion is severely calcified by visual estimation.
* Target lesion involves a bifurcation that requires intervention (usually, side branch >2 mm in diameter).
* Target lesion is totally occluded (100% stenosis usually associated with TIMI flow ≤1).
* Angiographic presence of probable or definite thrombus.
* Target vessel will be pre-treated with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon or transluminal extraction catheter prior to stent placement.
* Prior coronary intervention using brachytherapy to any segment of the target vessel.
* Angiographic restenosis of any segment of the target vessel that has undergone prior percutaneous coronary intervention.
* Angiographic evidence of atherosclerotic disease with > 50% diameter stenosis (by visual estimate) proximal or distal to the target lesion
* Prior surgical revascularization of the target vessel with a documented patent graft (either a saphenous vein or an arterial conduit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Vermeersch, MD, PhD, Principal Investigator — ZNA Middelheim, Department Interventional Cardiology; Maarten J. Suttorp, MD, PhD, Principal Investigator — St. Antonius Hospital

REFERENCES:
- [Result] Vermeersch P, Appelman Y, Horstkotte D, Richardt G, Boland J, Lalmand J, Coussement P, Castadot M, Janssens L, Agostoni P, Buysschaert I, Suttorp MJ. Safety and efficacy of the cobalt chromium PRO-Kinetik coronary stent system: results of the MULTIBENE study. Cardiovasc Revasc Med. 2012 Nov-Dec;13(6):316-20. doi: 10.1016/j.carrev.2012.09.006. PMID 23164477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 202 patients at 10 European sites have been enrolled.
Pre-assignment Details: Not group assignment.
Groups:
- BMS Implantation: BMS implantation
Period: Overall Study
Arm/Group | BMS Implantation
Started | 202 (5 patients with protocol violation were excluded.)
Completed | 197
Not Completed | 5
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Population: 197 patients were considered for baseline analysis. 5 patients with protocol violation were excluded.
Groups:
- BMS Implantation: Patients with a BMS implanted.
Arm/Group | BMS Implantation
Number analyzed (Participants) | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 97
  >=65 years | 100
Age Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 141
Region of Enrollment [Number; unit: participants]
  Belgium | 83
  Netherlands | 76
  Germany | 38

OUTCOME MEASURES:

1. Primary Outcome: Target Vessel Failure (TVF)
Description: Target vessel failure is defined as composite of revascularization, recurrent myocardial infarction, or cardiac death.
Time Frame: at 180 days post procedure
Population: Patients with follow up data available either 180 or 360 days post procedure.
Measure: Number; unit: participants
Arm/Group | BMS Implantation
Number analyzed (Participants) | 184
participants | 20

2. Secondary Outcome: Major Adverse Cardiac Events (MACE)
Description: MACE is defined as a composite of death, myocardial infarction, target lesion revascularization and coronary artery bypass grafting.
Time Frame: at 180 days post procedure
Population: Patients with follow up available either 180 or 360 days post procedure.
Measure: Number; unit: participants
Arm/Group | BMS Implantation
Number analyzed (Participants) | 184
participants | 21

ADVERSE EVENTS:
Arm/Group | BMS Implantation
Serious Adverse Events (participants affected / at risk) | 29/179
Other Adverse Events (participants affected / at risk) | 0/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS Implantation (N=179)
Target lesion revascularization (Cardiac disorders) | 20 (20)
Myocardial infarction (Cardiac disorders) | 3 (3)
Coronary artery bypass graft (Cardiac disorders) | 3 (3)
Cardiac death (Cardiac disorders) | 0 (0)
Non-cardiac death (General disorders) | 2 (2)
Target vessel revascularization (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations:

* missing comparators
* permission to conduct follow up visits by telephone
* limited number of 197 patients allows an insight of the safety and efficacy of the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less